CLINICAL TRIAL: NCT00354497
Title: Prostate Cancer Screening and Dietary HA Exposure in African-Americans: Phase II
Brief Title: Prostate Cancer Screening and Dietary Heterocyclic Amines in African American Men
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lawrence Livermore National Laboratory at University of California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Screening
Other Study IDs: CDR0000485428; LLNL-05-104
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2008-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Other: physiologic testing
Other: study of socioeconomic and demographic variables
Procedure: evaluation of cancer risk factors
Procedure: mutation carrier screening
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Screening may help doctors find prostate cancer sooner, when it may be easier to treat. The amount of heterocyclic amines in the diet may affect prostate cancer screening results and the risk of prostate cancer.

PURPOSE: This phase II trial is studying prostate cancer screening and dietary heterocyclic amines in African American men.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate dietary heterocyclic amine (HA) exposure in African American men who use HA-forming meats and cooking methods.
* Correlate dietary HA exposure with prostate-specific antigen and digital rectal exam screening results (i.e., higher HA exposure with increased abnormality in prostate cancer screening results) in these participants.

OUTLINE: This is a prospective study.

Participants complete a routine medical questionnaire and undergo a detailed dietary interview that focuses on meat consumption, cooking preferences, and other factors that may be associated with prostate cancer risk. Participants then undergo a digital rectal exam (DRE) and blood collection for prostate-specific antigen (PSA) testing (total PSA and % free PSA). Results of PSA testing and DRE, including follow-up instructions (if needed), are sent to the participant 3-4 weeks later.

Blood samples are also examined by phenotypic assays for UV-damage induced nucleotide excision-repair capacity.

PROJECTED ACCRUAL: A total of 800 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* African American male
* No previous diagnosis of prostate cancer
* Desires prostate cancer screening as a routine preventative medical service

PATIENT CHARACTERISTICS:

* Lives in or near Oakland, California
* Speaks English
* No medical or other disability (e.g., blindness, psychological dysfunction, or amputation) that would preclude study participation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2002-03

PRIMARY OUTCOMES:
Dietary heterocyclic amine (HA) exposure in African American men
Correlation of HA exposure with prostate cancer screening results

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth T. Bogen, DrPH, MPH, MA, ScD, Principal Investigator — Lawrence Livermore National Laboratory at University of California
Locations (2):
- United States (2):
  - Lawrence Livermore National Laboratory at University of California, Livermore, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California